CLINICAL TRIAL: NCT06921863
Title: Decisional Regret Following Radiotherapy Against Cancer With Poor to Excellent Prognosis
Brief Title: This Study Aims to Quantify Decisional Regret as Well as Quality of Life in Patients With Low- to High-risk Cancer and High Burden of Symptoms Undergoing Radiotherapy Using Established Questionnaires.
Acronym: DoItAgain
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Dr. med. Stephanie Bendrich, Dr. med. Stephanie Bendrich, University Medical Center Goettingen
Other Study IDs: 11/3/25
Record Dates: First submitted 2025-03-11; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Quality of Life (QOL); Decision Making ,Shared
Keywords: Decisional Regret; Radiotherapy; Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective registry study, patients with low-, intermediate- and high-risk tumor entities as well as patients with high symptom burden of any tumor entity in palliative constellation with indication for radiation treatment are included. This radiation treatment can be applied either as 3D-conformal RT or IGRT. The duration of treatment can range from one day to several weeks. For the primary endpoint as well as the secondary clinical and other exploratory endpoints, the 3 groups will be compared in terms of DR, QoL, toxicities and treatment plan parameters

DETAILED DESCRIPTION:
Decisional regret and quality of life are quantified and analyzed using general linear models (e.g. linear regression models, ANOVA), taking into account covariates such as tumor stage, application of further systemic therapies, extent of the radiation area, occurrence of acute and/or late side effects. Survival time analyses and tumor control rates are evaluated using Kaplan- Meyer and Cox regression. Technical endpoints, quality of life and patient satisfaction will be described descriptively and compared between the cohorts using a mixed linear model.

ELIGIBILITY:
Inclusion Criteria:

* Indication for radiotherapy
* Patient information and declaration of consent
* Patients age ≥ 18 years

Exclusion Criteria:

* previous radiotherapy in affected site or same localisation in group 1-3
* Inability to answer the questionnaires
* Pre-existing conditions with increased risk of acute or late toxicity (LiFraumeni, Crohn's disease, ulcerative colitis)
* Simultaneous participation in other studies that could interfere with this study and/or participation before expiry of a required restriction period
* Persons who are in a dependent/employment relationship with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Patients with low-risk cancers Cohort 2: Patients with cancers in the intermediate and high risk profile Cohort 3: Patients with high symptom burden
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Decisional Regret | from enrollment to the end of routinely performed clinical follow-up examinations after 5 yeasr after RT start
  Decisional Regret (DR) is measured by the German version of the Ottawa Decisional Regret Scale (Rühle et al. 2014) by answering the comprising 5 questions. Responses are provided on a five-point Likert scale. Decision regret is categorized as absent (0 points), mild (1-25 points) and strong (>25 points).
Quality of Life after Radiotherapy | from enrollment to the end of routinely performed clinical follow-up examinations after 5 yeasr after RT start
  Quality of Life is measured using the 80 question comprising PRO-CTCAE questionnaire version 1.0 (Hagelstein et al 2016) , the 30 question comprising EORTC QLQC30 questionnaire version 3.0 and the PSQ-18 questionnaire (Thayaparan and Mahdi 2013). All questionnaires have been previously validated in other publications.

IPD SHARING:
Plan to Share IPD: Undecided